CLINICAL TRIAL: NCT00384852
Title: A Phase 2, Multicenter, Double-Blind, Randomized, Stratified, Controlled, Efficacy, Safety and Feasibility Study of Recombinant Human Bone Morphogenetic Protein-2 (rhBMP-2)/Calcium Phosphate Matrix (CPM) as an Adjuvant Therapy in Closed Fractures of the Humerus
Brief Title: A Study of rhBMP-2/CPM in Closed Fractures of the Humerus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3100N7-212
Record Dates: First submitted 2006-10-03; First posted 2006-10-06 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Fractures
Keywords: Fracture; Humerus
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- A (Experimental): 1.0 mg/mL rhBMP-2/CPM + SOC
  Interventions: Drug: rhBMP-2/CPM
- B (Experimental): 2.0 mg/mL rhBMP-2/CPM + SOC
  Interventions: Drug: rhBMP-2/CPM
- C (Active Comparator): Buffer/CPM + SOC
  Interventions: Drug: rhBMP-2/CPM
- D (Other): Standard of Care Alone (SOC)
  Interventions: Drug: rhBMP-2/CPM

INTERVENTIONS:
Drug: rhBMP-2/CPM

SUMMARY:
The primary objective of this study is to assess whether fracture union is accelerated in subjects with humeral fractures (proximal,diaphyseal) treated with conservative therapy (standard of care) and a single dose of rhBMP-2/CPM compared to subjects who receive standard of care alone.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature subjects age 18 years or older.
* Subjects with either a closed proximal humeral fracture or a diaphyseal humeral fracture.
* Treatment plan that includes only conservative (nonoperative) therapy within 48 hours following injury.

Exclusion Criteria:

* Shoulder dislocation at the time of injury.
* Planned procedure(s) at that would stimulate fracture union at the time of application of the initial immobilization device.
* Fractures located in the distal third of humerus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2007-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable in this study is radiographic union. | Fracture union is assessed at 4, 6, 8, 10, 12, 16, 26 and 52 week visits. The goal of acceleration of fracture union will be met if median time to radiographic fracture union is decreased by 4 weeks in an active treatment arm compared to SOC alone.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Brazil, xavierl@wyeth.com; Trial Manager, Principal Investigator — For Mexico, gomezzlj@wyeth.com
Locations (34):
- United States (9):
  - Little Rock, Arkansas
  - Aurora, Colorado
  - Denver, Colorado
  - Clearwater, Florida
  - St. Petersburg, Florida
  - Brooklyn, New York
  - Monroe, North Carolina
  - Toledo, Ohio
  - State College, Pennsylvania
- Australia (3):
  - Herston, Queensland
  - Adelaide, South Australia
  - Melbourne, Victoria
- São Paulo, São Paulo, Brazil
- Canada (8):
  - Vancouver, British Columbia
  - Ajax, Ontario
  - Chatham, Ontario
  - Oshawa, Ontario
  - Scarborough Village, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Charlottetown
- Finland (2):
  - Oulu
  - Turku
- France (2):
  - Angers
  - Créteil
- Germany (2):
  - Berlin
  - Münster
- Mexico (4):
  - Chihuahua City, Chihuahua
  - Guadalajara, Jalisco
  - Monterrey, Nuevo León
  - D.f.
- Oslo, Norway
- Bucharest, Romania
- Linköping, Sweden

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196